CLINICAL TRIAL: NCT05137769
Title: Women's Responses to a Mindfulness-Based Body Scan: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Hannah G. Nolte, PhD Candidate, Principal Investigator, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 211345
Record Dates: First submitted 2021-11-15; First posted 2021-11-30 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Post Traumatic Stress Disorder; Trauma, Psychological
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Psychological Trauma | interventions — Whole Body Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Body Scan (Experimental): Participants will listen to a 20-minute, audio-guided mindfulness-based body scan exercise.
  Interventions: Behavioral: Body Scan

INTERVENTIONS:
Behavioral: Body Scan — The body scan is a core element of mindfulness-based stress reduction. Participants will listen to a 20-minute audio guide instructing them to focus on sensations in the body, place attention on one area of the body at a time, and progressively move attention throughout areas of the body.

SUMMARY:
PTSD develops after trauma and is marked by intrusive memories, avoidance of reminders, negative changes in mood and cognitive processes, and dysregulated physical and emotional stress reactivity. PTSD disparately affects twice as many women as men (8.0% vs. 4.1%), and finding effective treatments for these women is critical to reduce poor health outcomes associated with PTSD. Mind-body therapies (MBT), using the mind in combination with the body to facilitate healing hold promise to enhance PTSD treatment by improving stress regulation. While MBT reduce PTSD symptoms long-term, women with PTSD may initially experience distress, leading to treatment avoidance. This pilot study will explore women's initial responses to MBT, the prevalence of adverse responses, and which women are at risk for adverse responses in a sample of participants with a history of trauma and varying levels of PTSD symptoms. Study participants will attend one virtual study visit via one-on-one videoconference with the PI, where they will complete self-report measures of stress and affect before and after one session of a MBT exercise. A subset of the sample will complete a semi-structured individual videoconference interview with the PI within two weeks following completion of the MBT exercise and quantitative measures.

DETAILED DESCRIPTION:
The proposed single-group study will use a pre-post design to assess participants' responses to one exposure to a mindfulness-based body scan in a sample of women with a history of trauma and varying levels of PTSD symptoms. Quantitative measures will assess self-reported state positive affect, negative affect, and anxiety before and after the body scan, and psychosocial characteristics expected to influence responses. Individual semi-structured interviews will be conducted with a subsample of women to learn about their subjective experiences related to the body scan.

ELIGIBILITY:
Inclusion Criteria:

1. Previously experienced a traumatic event as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) >6 months prior,
2. self-identify as a woman and were assigned female sex at birth,
3. >18 years of age,
4. fluency in English,
5. access to computer or smartphone to complete REDCap surveys and videoconference study visit.

Exclusion Criteria:

1. active suicidal thoughts with a plan,
2. unable to abstain from drugs or alcohol for >48 hours prior to study videoconference,
3. current or history of psychosis with auditory and/or visual hallucinations,
4. meditated or practiced yoga >1 time(s) per month over past 6 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identify as a woman and were assigned female sex at birth
Enrollment: 60 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Positive Affect | Baseline to 1-minute post body scan
  Positive affect will be measured with The Positive and Negative Affect Schedule-Short Form (PANAS-SF), a 20-item questionnaire with 10 items assessing positive affect and 10 items assessing negative affect. Participants will be asked to "indicate to what extent you feel this way right now, that is, at the present moment" on a five-point scale; 1 = very slightly or not at all, 2 = a little, 3 = moderately, 4 = quite a bit and 5 = extremely. The positive affect score is obtained by adding the scores on items 1, 3, 5, 9, 10, 12, 14, 16, 17 and 19. The range of the possible total score is 10-50 with higher scores indicating greater positive affect.
Change in Negative Affect | Baseline to 1-minute post body scan
  Negative affect will be measured with The Positive and Negative Affect Schedule-Short Form (PANAS-SF), a 20-item questionnaire with 10 items assessing positive affect and 10 items assessing negative affect. Participants will be asked to "indicate to what extent you feel this way right now, that is, at the present moment" on a five-point scale; 1 = very slightly or not at all, 2 = a little, 3 = moderately, 4 = quite a bit and 5 = extremely. The negative affect score is obtained by adding the scores on items 2, 4, 6, 7, 8, 11, 13, 15, 18 and 20. The range of the possible scores is 10-50 with higher scores indicating greater negative affect.
Change in State Anxiety | Baseline to 1-minute post body scan
  State anxiety will be measured with The State-Trait Anxiety Inventory-State Form (STAI-S), a 20-item questionnaire with equal numbers of anxiety-present (e.g., "I feel tense") and anxiety-absent descriptors (e.g., "I feel calm"). Participants will be asked to indicate " how you feel right now, that is, at this moment" on a four-point scale; 1= not at all, 2 = somewhat, 3 = moderately so, 4= very much so. The anxiety-absent items (1, 2, 5, 8, 10, 11, 15, 16, 19, 20) will be reverse scored, and then all 20-items will be summed to obtain the state anxiety score. The range of the possible scores is 20-80; higher scores indicate greater state anxiety.
Participant Experience (qualitative) | 2 weeks post the in-person study visit.
  A subset of the sample (n=20) will complete a one-on-one telephone semi-structured interview to understand participant's perceived experience of the body scan exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah G Nolte, PhD(C), Principal Investigator — Vanderbilt University
Locations (4):
- United States (4):
  - Center of Hope, Columbia, Tennessee
  - Ascension Medical Group St Thomas Nashville, Nashville, Tennessee
  - Sterling Primary Care Associates - Centennial, Nashville, Tennessee
  - Empowered Heart, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No